CLINICAL TRIAL: NCT01204619
Title: Trial on Education And Clinical Outcomes for Home PD Patients (TEACH)
Acronym: TEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kook-Hwan Oh (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kook-Hwan Oh, Associate Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEACH
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Risk Reduction
Keywords: peritoneal dialysis
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional training group (No Intervention): in-center conventional training programs + two home visits
- Intensive training group (Experimental): in-center conventional training programs + an extra structured patient home visits repeatedly and regularly
  Interventions: Behavioral: Intensive training group

INTERVENTIONS:
Behavioral: Intensive training group — an extra structured patient centric training program on PD technique and diet according to the developed training curriculum
  Arms: Intensive training group

SUMMARY:
Since the emergence of home peritoneal dialysis as an alternative to in-center hemodialysis for chronic renal replacement therapy in the late 1970s, the percentage of dialysis patients on PD has continued to decrease each year. There have been a growing concern and research on patient and technique survival of peritoneal dialysis versus hemodialysis to find influential factors for better clinical outcomes. Meanwhile, technique failure rates were significantly higher in small centers treating less than twenty five PD patients. And there was a result for better technique survival after the second year, among the patients trained at the BREC(Baxter Renal Education Center). Better technique survival in large centers can be assumed with not only their more experience with patient management but also their educational infrastructure compared to small-sized centers.

Throughout our experiences in the last 30 years, we have recognized that a major element of PD program is patient training, however few data are available in terms of the relationship between PD training and treatment outcome and mostly are retrospective and non-randomized. Moreover, the technique survival and patient survival were analyzed with no significant difference.

From the insight, we decided to study prospectively to evaluate the efficacy of well-structured education program in terms of various patient outcomes in incident patients on PD.

DETAILED DESCRIPTION:
This study will be conducted as multi-center, open-label, randomized, controlled trial. One hundred four patient starting PD will be randomized into two training groups. Patients in the conventional training group (CG) will be given non-standardized in-center conventional training programs plus two sessions of training by home visit, while those in intensive training group (IG) given in-center conventional training programs plus repeated home visits regularly over 24-month period (total thirteen visits). The primary end point of the study is exit site infection (ESI). Secondary endpoints are peritonitis and all-cause infection. Generalized Estimating Equations will be used to assess the adjusted effect of training level on the ESI and Cox regression model employed to evaluate the effect on the peritonitis and other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Incident patients who have PD catheter insertion for starting PD with Baxter solutions
* > 20 yr of age

Exclusion Criteria:

* Patients who have undergone dialysis or received kidney transplant (note, however, that patients who are currently undergoing emergency hemodialysis temporarily right before the PD do not fall under the exclusion criteria.)
* Patients who are likely to receive kidney transplant or shift to hemodialysis within the following 1 year
* Patients diagnosed with acute inflammatory disease for the past three months
* Patients currently diagnosed with chronic inflammatory disease
* Currently pregnant or breastfeeding
* Patients who are involved in other clinical trial within 30 days prior to enrollment
* Patients who are currently hospitalized in care facilities such as nursing home, etc., or those who are expected to be hospitalized for the duration of the clinical test
* Patients who cannot perform PD by themselves
* Patients considered by the person in charge of the clinical test to have difficulty in participating in this clinical test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Exit site infection | 24 months

SECONDARY OUTCOMES:
time to the first peritonitis | 24 months
Number of ESIs per patient-month | 24 months
Days of hospitalization per year | 24 months
Systolic pressure and diastolic pressure measured at every visit | 24 months
Average number of antihypertensive medications | 24 months
Kt/V | 24 months
Residual renal function | 24 months
Fluid balance score | 24 months
Patient survival rate | 24 months
Total medical cost | 24 months
Total hours of education and training | 24 months
Unplanned home visit and education by peritoneal dialysis nurse | 24 months
Compliance score of patients | 24 months
HbA1c only for patients with diabetes | 24 months
Intact PTH level | 24 months
Hemoglobin level | 24 months
nPNA | 24 months
QOL | 24 months
SGA | 24 months
K level | 24 months
Total number of hospitalizations by cause over the last 1 and/or 2 years after the dialysis | 24 months
Technical survival rate | 24 months
peritonitis rate | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kook-Hwan Oh, M.D., PhD, Principal Investigator — Seoul National University
Locations (6):
- South Korea (6):
  - Wonkwang University, Sanbon Medical Center, Gunpo, Gyeonggi-do
  - Hallym University Sacred Hospital Puyngchon, Anyang
  - Gachon University Gil Hospital, Incheon
  - Eulji Medical Center, Seoul
  - Hallym University Sacred Hospital Gangdong, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No